CLINICAL TRIAL: NCT01025076
Title: Phase II Study of Evaluation of the Safety and Effectiveness of Stomaphyx for Transoral Incisionless Reduction of the Enlarged Gastric Pouch and Stoma
Brief Title: Evaluation of the Safety and Effectiveness of Stomaphyx for Transoral Incisionless Reduction of the Enlarged Gastric Pouch and Stoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Shahzeer Karmali, BSc, MD, FRCSC, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008913
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Morbid Obesity
Keywords: Enlarged gastric pouch and stoma; Post bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- StomaphyX Group (Experimental): * Primary Roux-en-Y gastric bypass with evidence of enlarged gastric pouch volume or enlarged stoma diameter of ≥ 20 mm via endoscopy or fluoroscopy.
  * Patients also demonstrate a weight regain of 15% of excess body weight loss.
  Interventions: Device: StomaphyX

INTERVENTIONS:
Device: StomaphyX — StomaphyX with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) is a transoral incisionless fastening device that allows for GI tissue approximation and creation of full-thickness (serosa-to-serosa) plications.

SUMMARY:
Executive Summary

Aims and Hypotheses of the Study:

The aim of the study will be to evaluate the safety, effectiveness and early outcome of the StomaphyX procedure for reducing the enlarged gastric pouch and stoma in post-bariatric patients. The study will test a hypothesis that the StomaphyX procedure will be effective in promoting the loss of regained weight, reducing the risk for comorbidities and improving patients' quality of life.

Type of Study: Prospective non-randomized Study Duration: 12 months Number of Patients: 20

Inclusion Criteria:

18-70 years of age, BMI ≥ 35, ≥ 2 years after primary Roux-en-Y gastric bypass with evidence of enlarged gastric pouch volume or enlarged stoma diameter of ≥ 20 mm via endoscopy or fluoroscopy. Pts also demonstrate a weight regain of 15% of excess body weight loss.

Exclusion Criteria:

Esophageal stricture, or any anatomic conditions that preclude passage of transoral endoluminal instruments, has another causal factor for weight regain other than stoma or pouch dilatation, portal hypertension, coagulation disorders or chronic use of anticoagulants, any active medical condition that would preclude the patient from completing the study or would result in an unreasonable risk to the patient.

Intervention Treatment: Creation of multiple full-thickness plications within the gastric pouch using the StomaphyX device (EndoGastric Solutions, Inc., Redmond, WA, USA)

Evaluation Criteria Primary Outcome: Change in body weight at 6 and 12 months Secondary Outcome: Gastric pouch volume assessment, stoma diameter determination, quality of life scores, waist circumference, co-morbidity resolution Effectiveness and Safety Assessment Clinical: Weight, height, waist circumference quality of life questionnaires (Impact of Weight QOL-Lite, Eating and Weight Patterns, Three-factor Eating, Emotional Eating Scale, GI QoL, GSRS and/or PGWB) Anatomical: Upper GI endoscopy, computed tomography or barium radiography Biochemical: Blood and urine tests (glucose, cholesterol, triglyceride, HDL, LDL, uric acid) Safety: Adverse events, complications, co-morbidities, hospital stay

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* BMI 35 or greater with one or more comorbidities
* At least 2 years post-Roux-en-Y gastric bypass surgery
* At enrollment, has regained at least 15% of excess body weight loss
* Enlarged Stoma Diameter
* Enlarged gastric pouch
* Completed successful nutritional screening and compliant with nutritional programs
* Completed successful cardiopulmonary evaluation
* Patient willing to cooperate with follow-up assessment tests
* Signed informed consent

Exclusion Criteria:

* Esophageal stricture or any anatomic conditions that preclude passage of transoral endoluminal instruments
* Has another causal factor for weight regain other than stoma or pouch dilatation such as non compliant with nutritional and exercise programs
* Portal hypertension
* Coagulation disorders or chronic use of anticoagulants
* Any active medical condition that would preclude the patient from completing the study or would result in an unreasonable risk to the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CAMIS, Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Thompson CC, Slattery J, Bundga ME, Lautz DB. Peroral endoscopic reduction of dilated gastrojejunal anastomosis after Roux-en-Y gastric bypass: a possible new option for patients with weight regain. Surg Endosc. 2006 Nov;20(11):1744-8. doi: 10.1007/s00464-006-0045-0. Epub 2006 Oct 5. PMID 17024527
- [Background] Elder KA, Wolfe BM. Bariatric surgery: a review of procedures and outcomes. Gastroenterology. 2007 May;132(6):2253-71. doi: 10.1053/j.gastro.2007.03.057. PMID 17498516
- [Background] Fernandez AZ Jr, DeMaria EJ, Tichansky DS, Kellum JM, Wolfe LG, Meador J, Sugerman HJ. Experience with over 3,000 open and laparoscopic bariatric procedures: multivariate analysis of factors related to leak and resultant mortality. Surg Endosc. 2004 Feb;18(2):193-7. doi: 10.1007/s00464-003-8926-y. Epub 2003 Dec 29. PMID 14691697
- [Background] Higa KD, Boone KB, Ho T. Complications of the laparoscopic Roux-en-Y gastric bypass: 1,040 patients--what have we learned? Obes Surg. 2000 Dec;10(6):509-13. doi: 10.1381/096089200321593706. PMID 11175957
- [Background] Sugerman HJ. Bariatric surgery for severe obesity. J Assoc Acad Minor Phys. 2001 Jul;12(3):129-36. PMID 11851201
- [Background] Gould JC, Garren MJ, Starling JR. Lessons learned from the first 100 cases in a new minimally invasive bariatric surgery program. Obes Surg. 2004 May;14(5):618-25. doi: 10.1381/096089204323093381. PMID 15186628
- [Background] Higa KD, Boone K, Nimeri A, Tercero F, Jackson A, Khan A. Gastric bypass: increased restriction for poor weight loss. Surg Endosc. 2007 Nov;21(11):1922-3. doi: 10.1007/s00464-007-9540-1. No abstract available. PMID 17909900
- [Background] Kaplan LM, Klein S, Boden G, Brenner DA, Gostout CJ, Lavine JE, Popkin BM, Schirmer BD, Seeley RJ, Yanovski SZ, Cominelli F. Report of the American Gastroenterological Association (AGA) Institute Obesity Task Force. Gastroenterology. 2007 May;132(6):2272-5. doi: 10.1053/j.gastro.2007.03.061. No abstract available. PMID 17498517
- [Background] Overcash WT. Natural orifice surgery (NOS) using StomaphyX for repair of gastric leaks after bariatric revisions. Obes Surg. 2008 Jul;18(7):882-5. doi: 10.1007/s11695-008-9452-8. Epub 2008 Apr 26. PMID 18438622
- [Background] Cadiere GB, Buset M, Muls V, Rajan A, Rosch T, Eckardt AJ, Weerts J, Bastens B, Costamagna G, Marchese M, Louis H, Mana F, Sermon F, Gawlicka AK, Daniel MA, Deviere J. Antireflux transoral incisionless fundoplication using EsophyX: 12-month results of a prospective multicenter study. World J Surg. 2008 Aug;32(8):1676-88. doi: 10.1007/s00268-008-9594-9. PMID 18443855
- [Background] Cadiere GB, Rajan A, Germay O, Himpens J. Endoluminal fundoplication by a transoral device for the treatment of GERD: A feasibility study. Surg Endosc. 2008 Feb;22(2):333-42. doi: 10.1007/s00464-007-9618-9. Epub 2007 Dec 11. PMID 18071818
- [Background] Cadiere GB, Rajan A, Rqibate M, Germay O, Dapri G, Himpens J, Gawlicka AK. Endoluminal fundoplication (ELF)--evolution of EsophyX, a new surgical device for transoral surgery. Minim Invasive Ther Allied Technol. 2006;15(6):348-55. doi: 10.1080/13645700601040024. PMID 17190659
- [Background] Jobe BA, O'Rourke RW, McMahon BP, Gravesen F, Lorenzo C, Hunter JG, Bronner M, Kraemer SJ. Transoral endoscopic fundoplication in the treatment of gastroesophageal reflux disease: the anatomic and physiologic basis for reconstruction of the esophagogastric junction using a novel device. Ann Surg. 2008 Jul;248(1):69-76. doi: 10.1097/SLA.0b013e31817c9630. PMID 18580209
- [Background] Deitel M, Gawdat K, Melissas J. Reporting weight loss 2007. Obes Surg. 2007 May;17(5):565-8. doi: 10.1007/s11695-007-9116-0. No abstract available. PMID 17658011
- [Background] Kolotkin RL, Crosby RD, Kosloski KD, Williams GR. Development of a brief measure to assess quality of life in obesity. Obes Res. 2001 Feb;9(2):102-11. doi: 10.1038/oby.2001.13. PMID 11316344
- [Background] Belle SH, Berk PD, Courcoulas AP, Flum DR, Miles CW, Mitchell JE, Pories WJ, Wolfe BM, Yanovski SZ; Longitudinal Assessment of Bariatric Surgery Consortium Writing Group. Safety and efficacy of bariatric surgery: Longitudinal Assessment of Bariatric Surgery. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):116-26. doi: 10.1016/j.soard.2007.01.006. PMID 17386392
- [Background] de Lauzon B, Romon M, Deschamps V, Lafay L, Borys JM, Karlsson J, Ducimetiere P, Charles MA; Fleurbaix Laventie Ville Sante Study Group. The Three-Factor Eating Questionnaire-R18 is able to distinguish among different eating patterns in a general population. J Nutr. 2004 Sep;134(9):2372-80. doi: 10.1093/jn/134.9.2372. PMID 15333731
- [Background] Karlsson J, Persson LO, Sjostrom L, Sullivan M. Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. Int J Obes Relat Metab Disord. 2000 Dec;24(12):1715-25. doi: 10.1038/sj.ijo.0801442. PMID 11126230
- [Background] Arnow B, Kenardy J, Agras WS. The Emotional Eating Scale: the development of a measure to assess coping with negative affect by eating. Int J Eat Disord. 1995 Jul;18(1):79-90. doi: 10.1002/1098-108x(199507)18:13.0.co;2-v. PMID 7670446
- [Background] Junghard O, Wiklund I. Validation of a four-graded scale for severity of heartburn in patients with symptoms of gastroesophageal reflux disease. Value Health. 2008 Jul-Aug;11(4):765-70. doi: 10.1111/j.1524-4733.2007.00313.x. Epub 2008 Jan 8. PMID 18194395
- [Background] Kulich KR, Madisch A, Pacini F, Pique JM, Regula J, Van Rensburg CJ, Ujszaszy L, Carlsson J, Halling K, Wiklund IK. Reliability and validity of the Gastrointestinal Symptom Rating Scale (GSRS) and Quality of Life in Reflux and Dyspepsia (QOLRAD) questionnaire in dyspepsia: a six-country study. Health Qual Life Outcomes. 2008 Jan 31;6:12. doi: 10.1186/1477-7525-6-12. PMID 18237386
- [Background] Matza LS, Boye KS, Yurgin N. Validation of two generic patient-reported outcome measures in patients with type 2 diabetes. Health Qual Life Outcomes. 2007 Jul 31;5:47. doi: 10.1186/1477-7525-5-47. PMID 17672906
- [Background] De Cocker KA, De Bourdeaudhuij IM, Cardon GM. What do pedometer counts represent? A comparison between pedometer data and data from four different questionnaires. Public Health Nutr. 2009 Jan;12(1):74-81. doi: 10.1017/S1368980008001973. Epub 2008 Mar 20. PMID 18353199

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | StomaphX
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- StomaphX: Patients with weight gain following VBG had endoluminal pouch reduction performed using the StomaphyXTM device in revisional bariatric surgery clinic
Arm/Group | StomaphX
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 1
Pre-operative weight [Mean (Standard Deviation); unit: Kg] | 119.5 (25.9)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Change in Body Weight
Description: Body weight changes at 6 months after StomaphyX procedure comparing to baseline weight.
Time Frame: At 6 months comparing to baseline weight
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | StomaphX
Number analyzed (Participants) | 14
kg | 9.6 (7.9)

ADVERSE EVENTS:
Arm/Group | StomaphX
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StomaphX (N=14)
headache (Surgical and medical procedures) | 2 (2)
low back pain (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No